CLINICAL TRIAL: NCT01732965
Title: Prospective Open Parallel Right to Left Bilateral Study Comparing Narrowband Ultraviolet B Alone Versus Narrowband Ultraviolet B and Psoralen Plus Ultraviolet A for the Treatment of Vitiligo
Brief Title: NB-UVB and PUVA Vitiligo Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Senior Staff Physician, Henry Ford Health System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFHS Vitiligo Phototherapy
Record Dates: First submitted 2012-11-13; First posted 2012-11-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Vitiligo
Keywords: Vitiligo; Phototherapy; Photochemotherapy
MeSH Terms: conditions — Vitiligo | interventions — Phototherapy; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NB-UVB phototherapy (Placebo Comparator): NB-UVB alone
  Interventions: Other: Phototherapy
- phototherapy and photochemotherapy (Experimental): NB-UVB and PUVA
  Interventions: Other: Phototherapy and Photochemotherapy

INTERVENTIONS:
Other: Phototherapy
  Arms: NB-UVB phototherapy
Other: Phototherapy and Photochemotherapy
  Arms: phototherapy and photochemotherapy

SUMMARY:
To evaluate if the combination of psoralen plus ultraviolet A and narrowband ultraviolet B is more effective than narrowband ultraviolet B alone in the treatment of vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Vitiligo affecting more than 15% body surface area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Determine the quantity of repigmentation | 6 months
  Determination the degree of repigmentation measured by the VASI score (Vitiligo area Scoring Index) after treating with the combination treatments (narrowband ultraviolet B and topical psoralen plus ultraviolet A) and compare it with narrowband ultraviolet B alone.

SECONDARY OUTCOMES:
Determine the quality of repigmentation. | Study initiation, 3 months and 6 months.
  Determination of the color of repigmentation, pattern of repigmentation, and the cessation of spread of vitiligo after treating with the combination treatments (narrowband ultraviolet B and topical psoralen plus ultraviolet A) and compare it with narrowband ultraviolet B alone.

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, MD, Principal Investigator — Henry Ford Dermatology
Locations (1):
- Henry Ford Dermatology, Detroit, Michigan, United States